### **Statistical Analysis Plan (SAP)**

Protocol Title: Oral ONC201 in Adult Recurrent Glioblastoma

Protocol Number: ONC006 (NCT02525692) Protocol Date: 03 June 2021 (Version 14.0) SAP Date: 24 May 2023 (Version 1.0)

# Statistical Analysis Plan

## ONC006

Oral ONC201 in Adult Recurrent Glioblastoma

I confirm that I have reviewed this document and agree with the content.

| | APPROVALS |
|---|---|
| Approved by: | Signature/Date: |
| Tom Brundage Vice President, Biostatistics Chimerix | DocuSigned by: \$\int \lambda \lambda \cdot \lambda \cdot \lambda \cdot \lambda \cdot \cdo |

## Table of Contents

| 1. | Introduction | 4 |
|----|---------------------|---|
| 2. | General Conventions | 4 |
| 3. | Analyses | 2 |

#### 1. Introduction

This abbreviated Statistical Analysis Plan (SAP) describes the statistical analyses to be conducted for the Study ONC006. For simplicity, reference is made to existing Integrated Summary of Safety (ISS) and Integrated Summary of Efficacy (ISE) SAPs when approaches are the same.

Study ONC006 is a Phase II, open-label, multi-center clinical trial of ONC201 in adult progressive/recurrent glioma with six arms. All subjects in Arm A receive oral ONC201 at 625 mg every 3 weeks and all subjects in Arms B, C, D, E, and F receive oral ONC201 at 625mg every week. Arms C and E include patients who have surgical resection of their tumor 1 day after the second (or more) dose of ONC201. All subjects remain on study until progressive disease, unacceptable toxicity or withdrawal of consent. For other study details, refer to the study protocol.

#### 2. General Conventions

The All Treated Analysis Set includes all patients who receive at least one dose of ONC201. This will be used for all analyses.

Unless otherwise specified, continuous variables will be summarized using descriptive statistics [number of observations, mean, standard deviation (SD), median, 1<sup>st</sup> (Q1) and 3<sup>rd</sup> (Q3) quartiles, minimum and maximum]. Categorical variables will be summarized as number (percent) of patients.

Day 1 is defined as the date of the first dose of study drug. For events that occur on or after Day 1, study day is defined as (date of event - date of Day 1 + 1). For events that occur prior to Day 1, study day is defined as (date of event - date of Day 1). There is no Day 0. Baseline is defined as the last observed measurement on or before the date of the first dose of study drug.

In general, other than for partial dates, missing data will not be imputed and will be treated as missing. Unless otherwise specified, partial dates will be imputed using the following rules:

- If year is missing, do not impute.
- If only day is missing, impute day as 1st of the month for start dates, end of the month for end dates, and 15<sup>th</sup> of the month for other dates.
- If day and month are missing, impute as January 1<sup>st</sup> for start dates, December 31<sup>st</sup> for end dates, and July 1<sup>st</sup> for other dates.

## 3. Analyses

All analyses will be presented by Arm and for All Patients. Otherwise, specified patient disposition, study drug usage, prior/concomitant/post-ONC201 medications, demographic and baseline characteristics, adverse events, and laboratories will use methods and summaries defined in the ISS SAP.

Laboratory boxplots will be presented for all tests with at least 60 patients having numeric baseline results: one plot per test, time on the x-axis, value on the y-axis. The plots will not be broken out by arm (i.e. only the All Patients group). Only Baseline and Cycles 2-12 will be presented. For Cycles 2-12, nominal visits will be used; if multiple values are associated with a visit, the highest value will be used for chemistry tests and lowest value will be used for hematology tests.

The following efficacy analyses will be performed: best overall response, overall response rate, disease control rate, duration of response, progression-free survival, and overall survival. All analyses will be

Chimerix, Inc. ONC006

based on the investigator-assessed overall RANO response. Discontinuation of treatment due to progressive disease will also be considered. All analyses, aside from overall survival, will be censored at the earlier of: (1) last disease assessment or (2) initiation of other anticancer therapy.

Cycle 1, 2 hour ONC201 plasma concentrations will be summarized descriptively.

Collected data contributing to presented tables and figures will be listed.

Other analyses specified in the protocol will either not be completed, or will be defined outside the scope of this plan.

Following is a complete list of the tables, figures, and listings to be prepared (with clarifying notes in parentheses).

| Number | Description |
|---|---|
| Table 1.1 | Patient Disposition |
| Table 1.2 | Demographics and Baseline Characteristics |
| Table 1.3 | Study Drug Usage |
| Table 1.4.1 | Prior Medications |
| Table 1.4.2 | Concomitant Medications |
| Table 1.4.3 | Post-ONC201 Medications |
| Table/Figure 2.1 | Progression-free Survival |
| Table/Figure 2.2 | Overall Survival |
| Table 2.3 | Response Rate (includes ORR, BOR, and DCR) |
| Table/Figure 2.4 | Duration of Response |
| Table 3.x.1* | Treatment-emergent Adverse Events (TEAE) |
| Table 3.x.2* | TEAE Grade 3 and Above |
| Table 3.x.3* | Serious TEAE |
| Table 3.x.4* | TEAE Leading to Death |
| Table 3.x.5* | TEAE Leading to Study Drug Discontinuation, Reduction, or Interruption |
| Table 3.x.6* | Study Drug Related TEAE |
| Table 3.x.7* | Study Drug Related TEAE Grade 3 and Above |
| Table 3.x.8* | Study Drug Related Serious TEAE |
| Table 3.x.9* | Study Drug Related TEAE Leading to Death |
| Table 3.x.10* | Study Drug Related TEAE Leading to Study Drug Discontinuation, Reduction, |
| | or Interruption |
| Table 3.x.11* | TEAE by Maxium Severity (overall only) |
| Table 3.x.12* | Study Drug Related TEAE by Maximum Severity (overall only) |
| Table 4.x.1* | Graded Laboratory Results (maximum post-baseline) |
| Table 4.x.2* | Graded Treatment-emergent Laboratory Results (maximum post-baseline, result |
| | only counted if > Baseline Grade) |
| Table 5.1 | Plasma Concentrations (Cycle 1, 2 hour only) |
| Figure 4.1 | Boxplot of Laboratory Results |
| Listing 1.1 | Patient Disposition |
| Listing 1.2 | Demographics and Baseline Characteristics |
| Listing 1.3 | Study Drug Usage |
| Listing 1.4 | Other Medications |
| Listing 2.1 | Efficacy Outcomes |
| Listing 3.1 | Adverse Events |
| Listing 3.2 | AE Leading to Death |
| Listing 3.3 | AE Leading to Study Drug Discontinuation, Reduction, or Interruption |
| Listing 4.1 | Listing of Graded Laboratory Results (includes all results for a patient/test where |
| | at least one post-baseline result is $\geq$ Grade 1) |
| Listing 5.1 | Plasma Concentrations (Cycle 1, 2 hour only) |
| x=1: all post-baselin | ne, x=2: prior to initiation of other anticancer therapy |